CLINICAL TRIAL: NCT04388436
Title: Cardiopulmonary and Immunological Impacts of Covid-19 in a Cohort of Survivors
Brief Title: Post Covid-19 Cardiopulmonary and Immunological Changes
Acronym: covid-19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: 20.05.67
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: COVID
Keywords: covid-19 cardiopulmonary immunological impact

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study rationale and aim: Resolving the COVID-19 pandemic quickly hinges on a crucial factor: how well a person's immune system remembers SARS-CoV-2, the virus behind the disease, after an infection has resolved and the patient is back in good health. This phenomenon, called immune memory, helps our bodies avoid reinfection by a bug persons have had before and influences the potency of life-saving treatments and vaccines. Also, the new coronavirus causes cardiac and pulmonary inflammation. So, our study planned to measure the cardiopulmonary and immunological changes in treated COVID-19 patients. Specific objectives: Measurement the duration of existence of COVID-19 IgM and IgG antibody in patient's plasma, detection of cardiac changes, pulmonary radiological and functional changes after COVID-19 infection. This could help detection of functional impairment in COVID-19 survivors which may have economic and social impact. Also, investigator will assess possible protective immune response following infection which may affect vaccination schedule. Methods: One hundred RT- PCR positive COVID-19 patients will be enrolled. HRCT chest, lateral flow immunoassay, spirometry, DLCO and Echo will be done on after 3, 6 and 12 months of discharge.

DETAILED DESCRIPTION:
• Background and significance:

COVID-19 (Coronavirus Disease-2019) is a public health emergency of international concern. Radiological, lung function changes were reported in different studies of pulmonary viral infection.

After a patient has recovered from severe acute respiratory syndrome (SARS), CT shows transient interlobular septal thickening and reticulation over a course of several weeks to months. The reticulation appears after the 2nd week and peaks around the 4th week. One-third of patients with persistent respiratory symptoms will have imaging findings of fibrosis, including interlobular and intralobular reticulation, traction bronchiectasis, and, rarely, honeycombing. Areas of air trapping, caused by damage to ciliated respiratory epithelium, have been reported in 92% of patients who have recovered from pneumonia and are less likely to resolve completely. Likewise, in patients with MERS, although the majority fully recover, 33% show evidence of lung fibrosis on follow-up imaging. These patients were commonly older, had prolonged ICU admission, and had greater lung involvement in the acute phase of the disease.

CT was performed 1 year after MERS-CoV infection in 65 (89%) patients. Radiological sequelae were revealed in 25% (4/16), 63% (19/30), and 95% (18/19) of patients in the no, mild, and severe pneumonia groups, respectively (P < 0.001). The median radiological sequelae score was 0, 1, and 3 in the no, mild, and severe pneumonia groups, respectively, and the radiological sequelae scores were significantly correlated with the severity of pneumonia (P < 0.001). The finding that more severe MERS pneumonia resulted in more impaired lung function strongly suggests that pulmonary sequelae can remain at least 1 year after MERS-CoV pneumonia, which is also supported by the correlation of radiological sequela correlated with the severity of MERS pneumonia.

A previous study showed that 24% of SARS survivors have impaired DLCO and 5% reduced lung volume at 12 months.

A follow-up study of 55 patients with SARS at 24 months revealed that 10 (18.2%), 9 (16.4%), 6 (10.9%) and 29 (52.7%) subjects had FEV1, FVC, TLC and DL(CO) < 80% of predicted values, respectively. The mean (SD) 6MWD increased significantly from 439.0 (89.1) m at 3 months to 460.1 (102.8) m at 6 months (P 0.016) and became steady after 6 months. However, 6MWD and 36 item Short Form General Health Survey scores were lower than the normal population throughout the study.

Pulmonary function defects were detected in half of the recovered severe acute respiratory syndrome patients 3 months after hospital discharge, but the impairment was mild in almost all cases. Many patients had reduced exercise capacity that cannot be accounted for by impairment of pulmonary function.

The deleterious SARS-CoV-2 infection myocardial effects could also be perpetuated by the prompt and severe downregulation of myocardial and pulmonary ACE2 pathways, thereby mediating myocardial inflammation, lung edema, and acute respiratory failure. ACE2 is widely expressed not only in the lungs but also in the cardiovascular system and, therefore, ACE2-related signalling pathways might even have a role in heart injury. Other proposed mechanisms of myocardial injury include a cytokine storm triggered by an imbalanced response by type 1 and 2 T-helper cells strong interferon-mediated immunopathological events and respiratory dysfunction and hypoxemia caused by COVID-19, resulting in damage to myocardial cells.

Infection due to viral, bacterial, or fungal pathogens initiates complex systemic inflammatory responses as part of innate immunity. Activation of host defense systems results in subsequent activation of coagulation and thrombin generation as critical communication components among humoral and cellular amplification pathways, a term called thromboinflammation or immunothrombosis.

Several serological immunoassays have been developed for the detection of SARS-CoV-2 viral proteins and antibodies in the serum or plasma. The most widely used biomarkers for the detection of SARS-CoV-2 infection in commercial immunoassays are IgM and IgG antibodies produced in suspects from the 2nd week of viral infection. IgM can be detected in the patient samples from 10 to 30 days after SARS-CoV-2 infection, while IgG can be detected from 20 days onwards. The IgM response occurs earlier than that of IgG, but it then decreases and disappears. On the other hand, IgG can persist after infection for a long time and may have a protective role.

A study reported that ELISA detected SARS-CoV-2 IgM or IgG in 34/40 individuals with an RT-PCR-confirmed diagnosis of SARS-CoV-2 infection (sensitivity 85%, 95%CI 70-94%), vs 0/50 pre-pandemic controls (specificity 100% [95%CI 93-100%]). IgG levels were detected in 31/31 RT-PCR positive individuals tested ≥10 days after symptom onset (sensitivity 100%, 95%CI 89-100%). IgG titres rose during the 3 weeks post symptom onset and began to fall by 8 weeks, but remained above the detection threshold. Point estimates for the sensitivity of lateral flow immunoassay (LFIA) devices ranged from 55-70% versus RT-PCR and 65-85% versus ELISA, with specificity 95-100% and 93-100% respectively.

• Timeliness, innovative nature and relevance of the project

AS COVID -19 is an emerging pandemic since late 2019, follow up studies of its sequelae are still lacking. The aim is to track any consequences regarding radiological findings, functional impairment of respiratory system and immunological response to COVID -19. This may have an economic and social burden if lung functions are deteriorating post infection. Also, development of an effective vaccination is an issue of great interest all over the world. Existence and duration of persistence of protective antibodies may help prediction of vaccination frequency and better understanding of the nature of the virus.

• Research design and methodologies:

One hundred RT- PCR positive COVID-19 patients will be enrolled.

The following data will be collected:

* Medical history: age, sex, occupation, comorbidities, previous treatment, …
* Clinical classification of COVID-19 infection:

  1- Mild: clinical symptoms without pneumonia 2- Moderate: clinical symptoms with pneumonia 3- Severe: who meet any of the following: respiratory rate 30 breath\minute, oxygen saturation less than 93% at rest and patient with more than 50%lesion progression within 24 to 48h in the lung
* Radiological data:

Pulmonary CT pattern of COVID-19 using Philips Ingenuity core 128 the Netherlands:

1. COVID-19 pneumonia, Type L:

   Only ground-glass densities are present on CT scan, primarily located subpleural and along the lung fissures. Consequently, lung weight is only moderately increased.
2. COVID-19 pneumonia, Type H:

The increased amount of non-aerated tissue Follow up CT at 3, 6 and 12 months intervals

Echocardiography using Sonoscape A5 portable echocardigraph:

3, 6 and 12 months intervals after clinical improvement

• Pulmonary function test: Spirometry: measurement of lung volumes and capacities (forced expiratory volume in first second FEV1, forced vital capacity FVC, FEV1\FVC and FEF25\75) Diffusion capacity of the lung to carbon monoxide (DLCO) at 3, 6 and 12 months intervals after clinical improvement

• Immunological data: Detection of COVID-19 IgG and IgM antibody in patient's plasma During infection and at 3, 6 and 12 months intervals after clinical improvement by BIOCREDIT COVID-19 IgG+ IgM Duo (One Step SARS-CoV-2 IgG and IgM Antibody Rapid Test) RapiGEN.INC.

BIOCREDIT COVID-19 IgG+ IgM Duo is a lateral flow immunochromatographic assay for qualitative detection of IgG and IgM specific to SARS-COV-2 virus in human serum, plasma and whole blood. Antihuman IgG and IgM conjugated with colloidal gold particles will react specifically with the SARS-COV-2 IgG and IgM antibodies in patient's serum, plasma and whole blood. The colloidal gold conjugated anti-human IgG & IgM and SARS-COV-2 specific IgG & IgM forms antibody-antibody-gold particle complex then it moves to pre-coated SARS-COV-2 NP and Spike protein recombinant antigens on the membrane. The reaction forms antigen-antibody-antibody-gold particle complex then they show as color band at T- line area. The control line (C) is used for procedural control and should always appear if the test is performed correctly.

• Detailed time plan

On discharge from hospital 1 month post discharge 3 months post discharge 6 months post discharge 12 months post discharge

CT angiographychest 1,3,6,12 months Lateral flow immunoassay 1,3,6,12 months Spirometry 1,3,6,12 months DLCO 1,3,6,12 months Echo 1,3,6,12 months

• Quality of the research team

Research team members are quick thinker, eager to know more and more, have analytical mind, show Commitment, cooperative and have excellent written and verbal communication skills. Also, the team is well qualified and has several national and international publications.

* Independent thinking and major research achievements This project will help us to know the sequalae of post infection by covid 19, regarding the immunological impact and the persistence of antibodies in the blood of survivors, persistent symptom, pulmonary remote effects in these patients.
* Impact

This study is set out to detect functional impairment in COVID-19 survivors which may have economic and social impact. Also, investigator will assess possible protective immune response following infection which may affect vaccination schedule

•

ELIGIBILITY:
Inclusion Criteria:

* pcr positive for covid -19 who are survived

Exclusion Criteria:

* dead patient uncooperative

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: covid-19 pcr positive survivors
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-07-10 (Estimated); Study Completion 2021-10-10 (Estimated)

PRIMARY OUTCOMES:
measurement of pulmonary function changes either obstructive or restrictive also lung diffusion and if there is remaining interstitial fibrosis | 12 months
  pulmonary function include lung volumes in millimetre and lung capacities
measurement for cardiac function and ejection fraction changes and if there is changes in pulmonary artery pressure | 12 months
  Ejection fraction ,myocardial contractility,pulmonary artery pressure

SECONDARY OUTCOMES:
assessment of IGM and IGG level and if there is immunological changes | 12 months
  IGG,IGM level using rapid covid antibody titre

CONTACTS AND LOCATIONS:
Overall Officials: Tamer A Elhadidy, MD, Principal Investigator — assistant professor
Locations (1):
- Mansoura faculty of medicine, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
no plan for sharing data for other researchers

REFERENCES:
- [Background] Wong CK, Lam CW, Wu AK, Ip WK, Lee NL, Chan IH, Lit LC, Hui DS, Chan MH, Chung SS, Sung JJ. Plasma inflammatory cytokines and chemokines in severe acute respiratory syndrome. Clin Exp Immunol. 2004 Apr;136(1):95-103. doi: 10.1111/j.1365-2249.2004.02415.x. PMID 15030519
- [Background] Vashist SK. In Vitro Diagnostic Assays for COVID-19: Recent Advances and Emerging Trends. Diagnostics (Basel). 2020 Apr 5;10(4):202. doi: 10.3390/diagnostics10040202. PMID 32260471
- [Background] Park WB, Jun KI, Kim G, Choi JP, Rhee JY, Cheon S, Lee CH, Park JS, Kim Y, Joh JS, Chin BS, Choe PG, Bang JH, Park SW, Kim NJ, Lim DG, Kim YS, Oh MD, Shin HS. Correlation between Pneumonia Severity and Pulmonary Complications in Middle East Respiratory Syndrome. J Korean Med Sci. 2018 May 10;33(24):e169. doi: 10.3346/jkms.2018.33.e169. eCollection 2018 Jun 11. PMID 29892209
- [Background] Oudit GY, Kassiri Z, Jiang C, Liu PP, Poutanen SM, Penninger JM, Butany J. SARS-coronavirus modulation of myocardial ACE2 expression and inflammation in patients with SARS. Eur J Clin Invest. 2009 Jul;39(7):618-25. doi: 10.1111/j.1365-2362.2009.02153.x. Epub 2009 May 6. PMID 19453650
- [Background] Ooi GC, Khong PL, Muller NL, Yiu WC, Zhou LJ, Ho JC, Lam B, Nicolaou S, Tsang KW. Severe acute respiratory syndrome: temporal lung changes at thin-section CT in 30 patients. Radiology. 2004 Mar;230(3):836-44. doi: 10.1148/radiol.2303030853. PMID 14990845
- [Background] Ong KC, Ng AW, Lee LS, Kaw G, Kwek SK, Leow MK, Earnest A. 1-year pulmonary function and health status in survivors of severe acute respiratory syndrome. Chest. 2005 Sep;128(3):1393-400. doi: 10.1378/chest.128.3.1393. PMID 16162734
- [Background] Ngai JC, Ko FW, Ng SS, To KW, Tong M, Hui DS. The long-term impact of severe acute respiratory syndrome on pulmonary function, exercise capacity and health status. Respirology. 2010 Apr;15(3):543-50. doi: 10.1111/j.1440-1843.2010.01720.x. Epub 2010 Mar 19. PMID 20337995
- [Background] Jackson SP, Darbousset R, Schoenwaelder SM. Thromboinflammation: challenges of therapeutically targeting coagulation and other host defense mechanisms. Blood. 2019 Feb 28;133(9):906-918. doi: 10.1182/blood-2018-11-882993. Epub 2019 Jan 14. PMID 30642917
- [Background] Ketai L, Paul NS, Wong KT. Radiology of severe acute respiratory syndrome (SARS): the emerging pathologic-radiologic correlates of an emerging disease. J Thorac Imaging. 2006 Nov;21(4):276-83. doi: 10.1097/01.rti.0000213581.14225.f1. PMID 17110851
- [Background] Hui DS, Wong KT, Ko FW, Tam LS, Chan DP, Woo J, Sung JJ. The 1-year impact of severe acute respiratory syndrome on pulmonary function, exercise capacity, and quality of life in a cohort of survivors. Chest. 2005 Oct;128(4):2247-61. doi: 10.1378/chest.128.4.2247. PMID 16236881
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Engelmann B, Massberg S. Thrombosis as an intravascular effector of innate immunity. Nat Rev Immunol. 2013 Jan;13(1):34-45. doi: 10.1038/nri3345. Epub 2012 Dec 7. PMID 23222502
- [Background] Das KM, Lee EY, Singh R, Enani MA, Al Dossari K, Van Gorkom K, Larsson SG, Langer RD. Follow-up chest radiographic findings in patients with MERS-CoV after recovery. Indian J Radiol Imaging. 2017 Jul-Sep;27(3):342-349. doi: 10.4103/ijri.IJRI_469_16. PMID 29089687
- [Background] Cameron MJ, Bermejo-Martin JF, Danesh A, Muller MP, Kelvin DJ. Human immunopathogenesis of severe acute respiratory syndrome (SARS). Virus Res. 2008 Apr;133(1):13-9. doi: 10.1016/j.virusres.2007.02.014. Epub 2007 Mar 19. PMID 17374415
- See also: Viral kinetics and antibody responses in patients with COVID-19 — https://www.medrxiv.org/content/10.1101/2020.03.24.20042382v1.abstract
- See also: Antibody testing for COVID-19: A report from the National COVID Scientific Advisory Panel — https://www.medrxiv.org/content/10.1101/2020.04.15.20066407v2